CLINICAL TRIAL: NCT02410109
Title: Developing an Integrated Model for Home Visitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00071007; 1R34MH093514-01 (NIH)
Record Dates: First submitted 2012-03-15; First posted 2015-04-07 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCRIPT intervention (Experimental)
  Interventions: Behavioral: SCRIPT integrated model
- Historical Control (No Intervention)

INTERVENTIONS:
Behavioral: SCRIPT integrated model — Perinatal women will be screened for psychosocial risks at time of home visiting enrollment. Women exhibiting elevated depressive symptoms and/or have a history of clinical depression who are not currently clinically depressed will be referred for depression prevention services. Women experiencing a depressive episode will be referred for group CBT. Women who screen positive for elevated anxiety symptoms, PTSD symptoms, intimate partner violence, or substance abuse will be referred to a mental health or social service agencies. If a client is referred for services, the assessment worker will provide written educational materials about the risk factor that is being addressed through the referral. At the first home visit, the home visitor will discuss these educational materials.
  Arms: SCRIPT intervention

SUMMARY:
Perinatal depression is a significant concern, particularly for low-income women. Many cases of perinatal depression are complicated by comorbidities such as post-traumatic stress disorder symptoms, anxiety, and intimate partner violence. Providing perinatal mental health services to women in home visiting programs could have considerable public health significance. This study will develop and test an integrated model of mental health services embedded within home visitation (HV) programs. This model will (1) incorporate a protocol for systematic screening and referral; (2) strengthen formal linkages between HV programs and other components of service systems; (3) promote the capacity of service systems to provide evidence-based early intervention and treatment for depression; and (4) facilitate the receipt of early intervention and treatment services for perinatal depression and comorbid conditions. This will be the first model to our knowledge that systematically integrates screening, referral, and early intervention and treatment for perinatal depression and associated comorbidities within HV programs.

The specific aims are:

1. To develop an integrated model of perinatal depression care within HV programs. This integrated model ("SCRIPT") will incorporate screening, referral, and individualized prevention and treatment services.
2. To assess the feasibility of implementing the SCRIPT model with high fidelity in two HV programs. One HV program-DRUM Healthy Families-will use paraprofessionals as interventionists while the other program-M&I Nursing-will use nurses and social workers as interventionists.
3. To determine the impact of the SCRIPT model on depressive symptoms and major depressive episodes.

ELIGIBILITY:
Inclusion Criteria:

* pregnant or child < 6 months
* enrolled in Baltimore City home visiting program

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 178 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | Baseline, 3 months, 6 months
  Change in scores on the Beck Depression Inventory measured over 3 time points.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - DRUM Healthy Families, Baltimore, Maryland
  - Maternal and Infant Nursing Program, Baltimore, Maryland